CLINICAL TRIAL: NCT05473676
Title: Robotic Walking for Children Who Cannot Walk
Acronym: RoWaCaWa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Elizabeth Condliffe, PhD MD, Assistant Clinical Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB21-1166
Record Dates: First submitted 2022-04-22; First posted 2022-07-26 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy; Mobility Limitation; Brain Injuries; Spinal Cord Injuries; Spina Bifida
Keywords: Robot Assisted Gait Training; Trexo; Rehabilitation; Robotic Training; Assisted Walking
MeSH Terms: conditions — Cerebral Palsy; Mobility Limitation; Brain Injuries; Spinal Cord Injuries; Spinal Dysraphism

STUDY DESIGN:
Intervention Model Description: All participants will proceed through the same study timeline from the time of enrollment.
Masking Description: Because there is only 1 arm in the study, and each participant proceeds through the same study timeline, participants, care providers, investigators, and outcome assessors will know the intervention received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robotic Training Period (Experimental): Participants will engage in robot assisted gait training on at least 5 days/week for at least 30 minutes each day, for a total period of 12 weeks.
  Interventions: Device: Robotic Training Period

INTERVENTIONS:
Device: Robotic Training Period — Participants will engage in robot assisted gait training on at least 5 days/week for at least 30 minutes each day, for a total period of 12 weeks.

SUMMARY:
A common problem among children with nervous system disorders is difficulty walking on their own. This has impacts beyond mobility including short and long-term health conditions associated with physical inactivity and different developmental experiences as a result of the mobility impairments. A robotic trainer can both provide rehabilitation and be an assistive device to help compensate for difficulties. Figuring out how to prescribe it is critical to improve daily life for children with significant disabilities. Preliminary use of robotic trainers have shown many benefits, such as better head control and improved independence in transfers, which greatly increases ability to live independently. Additionally, vital functions that are frequently impaired in those with less physical activity, such as sleep and bowel habits, seem to improve. Finally, these children enjoy using them.

This project aims to determine who is most likely to benefit from training with a robotic trainer and investigate key details about the dose of training that is needed. Families that are already using or hope to use robotic training need this data to help improve their access to the intervention. Clinicians need this systematic approach to building evidence to ensure a future multi-centre randomized control trial is well designed. This study is needed to help improve the lives of those who live with significant disabilities. The objective is to evaluate the feasibility and impacts of delivering robotic gait training at home. Integral in this study is capturing the user perspectives. This will both provide preliminary evidence-based advice to potential users, their families, and clinicians as well as provide key metrics to design a definitive multi-centre randomized control trial.

The investigators will provide robotic gait trainers, specifically Trexo robotic gait trainers, to participants and their families to use in their home communities for 12 weeks to evaluate the feasibility and impacts of intensive robotic gait training in people who cannot walk independently. Assessments will be completed throughout the duration of study, including before, during, and after the training intervention, with the goal of evaluating a wide range of feasibility considerations and impacts from robotic training.

ELIGIBILITY:
Inclusion Criteria:

* At least 4 years of age
* Unable to walk independently due to pediatric onset, non-progressive central nervous system disorder or injury (ie. cerebral palsy or acquired brain injury)
* Able to fit into Trexo robotic gait trainer (both leg length and weight)
* Able to fulfill training requirements throughout training period (5 days/week for at least 30 minutes each session)
* Able to comply with study procedures (assessments, training)

Exclusion Criteria:

* Medical condition or recent surgery requiring lower extremity immobilization or weight-bearing restrictions (ie. fracture, unstable hip subluxation).
* Medical condition requiring a physical activity restriction (ie. unstable arrhythmia).
* Pain or symptomatic hypotension while standing.
* Contracture such that the Trexo robotic gait trainer does not result in forward movement.
* Current involvement in a potentially confounding intervention (determined on a case-by-case basis).

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Training Time | Assessed throughout the 12 weeks (Week 5 through Week 16) robotic training period.
  Time spent in the trainer each session, total time spent in the trainer (weekly, monthly).
Training Frequency | Assessed throughout the 12 week (Week 5 through Week 16) robotic training period.
  Frequency of training sessions (days/week).
Canadian Occupational Performance Measures (COPM) | Assessed at enrollment (Week 0), before Robotic Gait Training period (~Week 4), following Robotic Gait Training period (~Week 16), and at 3-months post-training (~Week 28).
  Structured questions and rating scales to determine problem areas and goals for training. Identified problems are scored on a 10 point scale, 1 being not able to complete the task at all.
Goal Attainment Scaling | Assessed at enrollment (Week 0), before Robotic Gait Training period (~Week 4), following Robotic Gait Training period (~Week 16), and at 3-months post-training (~Week 28).
  Rating of success in achieving an outcome or desired goal (identified using the COPM), where 0 = the expected level of achievement, -2 = much less achieved than expected, and +2 = much more achieved than expected.
Early Clinical Assessment of Balance (ECAB) | Assessed monthly from time of enrollment through 3-months post-training.
  Clinical balance assessment to determine participant's balance capabilities.

SECONDARY OUTCOMES:
Number of Participants Enrolled and Completed | Assessed throughout the study duration, an average of 7-9 months depending on time of enrollment..
  Assessment of number of participants that start the study and how many are able to complete the study.
Caregiver Priorities & Child Health Index of Life with Disabilities (CP-CHILD) | Assessed before (~Week 4) and after (~Week 16) robotic gait training.
  Qualitative assessment of impacts of robotic gait training on participants and families.
EQ-5D-Y (Youth) | Assessed before (~Week 4) and after (~Week 16) robotic gait training.
  Qualitative assessment of impacts of robotic gait training on participants and families.
CarerQOL | Assessed before (~Week 4) and after (~Week 16) robotic gait training.
  Qualitative assessment of impacts of robotic gait training on participants and families.
Focus Groups | Assessed before (~Week 4) and after (~Week 16) robotic gait training.
  Semi-structured interviews with participants and families and/or caregivers. Themes will include independence in daily function and feedback on training with the device.
Head Control While Walking | Assessed at enrollment (Week 0), before Robotic Training Period (~Week 4), after Robotic Training Period (~Week 16), and 3-months post-training (~Week 28)..
  Head angle from vertical will be measured to determine if head control is impacted by training.
Seated Limits of Stability | Assessed at enrollment (Week 0), before Robotic Training Period (~Week 4), after Robotic Training Period (~Week 16), and 3-months post-training (~Week 28).
  Forward, backward, and side to side leaning will be assessed to evaluate trunk strength and control.
Ramp & Hold | Assessed at enrollment (Week 0), before Robotic Training Period (~Week 4), after Robotic Training Period (~Week 16), and 3-months post-training (~Week 28).
  Evaluation of stiffness and involuntary muscle activity, recorded using electromyography (EMG) or mechanomyography (MMG).
Voluntary Muscle Activity | Assessed at enrollment (Week 0), before Robotic Training Period (~Week 4), after Robotic Training Period (~Week 16), and 3-months post-training (~Week 28).
  Evaluation of voluntary muscle contractions. Recorded using EMG or MMG.
Modified Tardieu Scale | Assessed monthly from time of enrollment (Week 0) through to 3-months post-training (~Week 28).
  Clinician movement of joint to determine range of motion and angle of catch at the joint. Joint neutral is defined as 0 degrees, where any range beyond neutral is recorded in "+" degrees and any range not reaching neutral is recorded in "-" degrees.
Habitual Activity Estimation Scale (HAES) | Assessed monthly from time of enrollment (Week 0) through to 3-months post-training (~Week 28).
  Participant or proxy report of estimated physical activity during a typical weekday and week-end day. Participants or proxy report a percentage of time spent inactive, somewhat inactive, somewhat active, and active on a typical weekday and week-end day.
PROMIS Sleep Disturbance Questionnaire | Assessed monthly from time of enrollment (Week 0) through to 3-months post-training (~Week 28).
  Participant or proxy report of sleep disturbances. Participants or a proxy will rate different sleep scenarios on a 5 point scale, 1 being Never and 5 being Always.
Heart Rate Reserve | Assessed continually for 1 week at Week 0, ~Week 4, ~Week 5-8 (once), ~Week 12-16 (once), ~Week 17, and ~Week 28
  Week-long assessment measuring heart rate, tracked using Actigraph wearable sensor worn on chest and wrist.
Distance Walked | Assessed continually for 1 week at Week 0, ~Week 4, ~Week 5-8 (once), ~Week 12-16 (once), ~Week 17, and ~Week 28
  Week-long assessment measuring heart rate, tracked using inertial measurement units (IMUs) worn on feet.
Sleep Duration | Assessed continually for 1 week at Week 0, ~Week 4, ~Week 5-8 (once), ~Week 12-16 (once), ~Week 17, and ~Week 28
  Week-long assessment measuring heart rate, tracked using Actigraph wearable sensor worn on chest and wrist.
Bowel Function | Assessed continually for 1 week at Week 0, ~Week 4, ~Week 5-8 (once), ~Week 12-16 (once), ~Week 17, and ~Week 28
  Week-long assessment measuring frequency and quality of bowel movements as well as any interventions used to facilitate bowel movements, for example medications. Tracked using participant or proxy reports in a daily diary provided by study team.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth G Condliffe, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Pediatric Onset of Neuromotor Impairments Lab, Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
There is an Open Science plan to share de-identified IPD. All data collected in this study will be de-identified and added to a robotic training database. Access by other researchers must be requested, and agree to a Terms of Use agreement before access is granted.
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available at the end of the study. There is no plan to close the database.
Access Criteria: Researchers requesting access to the database will be required to sing a Terms of Use agreement.